CLINICAL TRIAL: NCT06824025
Title: Comparison of Nebulized Neostigmine/Atropine Versus Lignocaine in Treating Acute Post-dural Puncture Headache Following Subarachnoid Block in Parturient Undergoing Elective Cesarean Section. A Randomized, Clinical Trial.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1392-12-2024
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Nebulization of 4 mL 0.9% saline twice daily for three days plus conventional management (consisted of bed rest in the supine position, good hydration with continuous infusion of 30 mL/kg/day lactated Ringer solution, 1 g paracetamol every 6 h. Diclofenac sodium suppository (100 mg) was given twice daily for 5 days as routine post-operative pain management
  Interventions: Drug: lidocaine group ( nebulized lidocaine + saline) total volume 4 ml
- Neostgmine group (Active Comparator): Nebulization of 20 µ/kg neostigmine and 10 µ/kg atropine diluted in 0.9% sterile saline ( total volume 4 ml) twice daily for three days plus conventional management ( consisted of bed rest in the supine position, good hydration with continuous infusion of 30 mL/kg/day lactated Ringer solution, 1 g paracetamol every 6 h. Diclofenac sodium suppository (100 mg) was given twice daily for 5 days as routine post-operative pain management
  Interventions: Drug: lidocaine group ( nebulized lidocaine + saline) total volume 4 ml
- Lidocaine group (Active Comparator): Nebulization of lidocaine 20% (60 mg) diluted in 4 ml of sterile saline 0.9% twice daily for three days plus conventional management ( consisted of bed rest in the supine position, good hydration with continuous infusion of 30 mL/kg/day lactated Ringer solution, 1 g paracetamol every 6 h. Diclofenac sodium suppository (100 mg) was given twice daily for 5 days as routine post-operative pain management
  Interventions: Drug: lidocaine group ( nebulized lidocaine + saline) total volume 4 ml

INTERVENTIONS:
Drug: lidocaine group ( nebulized lidocaine + saline) total volume 4 ml — nebulization of 60 mg lidocaine in 4ml saline 0.9%

SUMMARY:
Post-dural puncture headache (PDPH) is a common and debilitating complication of spinal anesthesia in pregnant patients undergoing cesarean sections, with an incidence ranging from 0.5% to 2% (1). The International Headache Society (IHS) defines PDPH as a headache occurring within 4 days of a lumbar puncture, caused by cerebrospinal fluid (CSF) leakage through the dural puncture (2). Although the exact cause of PDPH is not fully understood, it is thought to occur due to cerebrospinal fluid loss through dural tears, which leads to tension on pain-sensitive intracranial structures and reflex, uncontrolled cerebral vasodilation leading to severe agonizing tension headache (3). Treatment options include proper hydration, maintaining a supine position, caffeine, paracetamol, nonsteroidal anti-inflammatory drugs (NSAIDs). Many adjuvants have been questioned for their therapeutic effectiveness in enhancing conservative medical treatments, with conflicting results (4). For example, sumatriptan, theophylline and dexmedetomidine have been extensively studied. Neostigmine has emerged as a promising pharmacological adjuvant for conservative management. Neostigmine increases the serum level of acetylcholine via inhibition of cholinesterase (5). This action mediates cerebral vasoconstriction via nicotinic receptors, thus antagonizing the unopposed vasodilatation occurred due to dural tear. Lidocaine, on the other hand, can mediate sphenopalatine ganglion block which is responsible for pain signals transmission from the face (6).

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old parturient with post partum headache after elective CS under spinal anesthesia with visual analog score (VAS) ≥ 4 [14] and Lybecker classification score ≥ 2

Exclusion Criteria:

* Pregnancy induced hypertension
* Emergency C.S
* Asthmatic candidates
* Previous history of migraine or trigeminal neuralgia
* History of bronchial asthma
* Post partum hemorrhage
* Need for GA , failed spinal anesthesia
* Patient refusal

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
VAS score | 3 days
  Acute pain categorization. 10= severe umimaginable pain..... 7- 9= severe pain...4-6= moderate to severe pain ..3- 5= moderate pain .... 1-3= mild pain

SECONDARY OUTCOMES:
Lybecker headache | 72 hours
  Severity of headache . mild, moderate , severe headache
number of patients in need for epidural blood patch | 3 days
  VAS>3
procedure related complication | 3 days
  Complications related to nebulization ( dry cough, spasm, colics......)
neural complications | 7 days
  persistent neural complications at time of discharge
hospital stay | 7 days
  length of hospital stay
Trans-cranial doppler | at onset of treatment, 24, 72 hours
  Mean flow velocity
transcranial doppler | at enrollment, 24,72 hours
  resistive index